CLINICAL TRIAL: NCT05635487
Title: A Phase II Study of SHR-A1811 Monotherapy or Combined With Pyrotinib Maleate as Neoadjuvant Treatment in HER2-positive Breast Cancer Patients
Brief Title: A Study of SHR-A1811 Monotherapy or Combined With Pyrotinib Maleate as Neoadjuvant Treatment in HER2-positive Breast Cancer Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Caigang Liu, Director of the Cancer Center, Shengjing Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MUKDEN 07
Record Dates: First submitted 2022-11-15; First posted 2022-12-02 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: HER2-positive Breast Cancer
Keywords: SHR-A1811; Pyrotinib; HER2-positive Breast Cancer; Neoadjuvant
MeSH Terms: interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811+Pyrotinib (Experimental)
  Interventions: Drug: SHR-A1811; Drug: Pyrotinib
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811
Drug: Pyrotinib — Pyrotinib
  Arms: SHR-A1811+Pyrotinib

SUMMARY:
This is a phase II trial evaluating the efficacy and safety of SHR-A1811 monotherapy or combined with pyrotinib maleate in Stage II-III HER2-positive breast cancer. Subjects will receive the neoadjuvant therapy of SHR-A1811 monotherapy or combined with pyrotinib for six cycles, and then undergo surgery within 4 weeks after neoadjuvant therapy. Efficacy will be assessed every 2 cycles.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 but ≤ 75 years
* Histologically confirmed to be HER2-positive invasive breast cancer
* Treatment-naive patients with stage II-III
* Eastern Cooperative Oncology Group (ECOG) score 0-1
* Good level of organ function

Exclusion Criteria:

* Previously received any anti-tumor therapy (chemotherapy, radiotherapy, molecular targeted therapy, endocrine therapy, etc.)
* Received any other anti-tumor therapy at the same time
* Bilateral breast cancer, inflammatory breast cancer or occult breast cancer
* Stage IV breast cancer
* With a history of any malignancies in the past 5 years, excluding cured cervical carcinoma in situ and melanoma skin cancer
* Inability to swallow, chronic diarrhea, intestinal obstruction, and a variety of factors affecting drug administration and absorption
* Participated in other drug clinical trials within 4 weeks before enrollment
* History of allergies to the drug components of this protocol
* Clinically significant pulmonary diseases
* Clinically significant cardiovascular diseases
* History of immunodeficiency
* Active hepatitis and liver cirrhosis

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Total pathological complete response (tpCR: ypT0-is/ypN0) | At the time of surgery

SECONDARY OUTCOMES:
Breast pathological complete response (bpCR：ypT0-is) | At the time of surgery
Residual cancer burden (RCB) | At the time of surgery
Best overall response rate (BORR) | During 18 weeks of the neoadjuvant treatment
Overall survival (OS) | 5 years
Disease-free survival (DFS) | 5 years
Event-free survival (EFS) | 5 years
Health-related quality of life (HRQOL) (EORTC QLQ-C30) | During 18 weeks of the neoadjuvant treatment
  The European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ) Core 30 (EORTC QLQ-C30)
Health-related quality of life (HRQOL) | During 18 weeks of the neoadjuvant treatment
  The European Organization for Research and Treatment of Cancer (EORTC) quality of life questionnaire Breast Cancer (EORTC QLQ- BR23) will be used to measure the HRQOL.

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, MD, Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital affiliated to China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No